CLINICAL TRIAL: NCT06527651
Title: Effects of Ultrasound-guided Genicular Nerve Block in Knee Osteoarthritis Patients on Proprioception and Static Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2024-07-16; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Osteoarthritis; Osteoarthritis, Knee; Proprioceptive Disorders; Balance; Distorted
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Somatosensory Disorders | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genicular blocks (Other): Genicular blocks were applied bilaterally by another physiatrist who was experienced in ultrasonographic (US) interventional procedures more than 5 years. Total of 6mL solution consisting of 0.5 mg/2mL dexamethazone and 4mL %1 lidocaine for three branches of genicular nerves (superomedial, superolateral and inferomedial branches) was divided into three branches for each knee. Total of 12 mL solution was applied for each patient. Antiseptic precautions were taken, sterile environment was prepared. A 5-12 MHz linear probe (Loqiq P5, GE Medical systems) was used for all US evaluations. The probe was positioned in line with the femur shaft. Firstly to find the superomedial genicular nerve, probe was moved to the junction of femur shaft and medial femoral condyle. Color doppler was used to clarify superomedial genicular artery and 2mL injection solution was applied around the pulsatile artery region.
  Interventions: Drug: Genicular blocks (dexamethazone and lidocaine)

INTERVENTIONS:
Drug: Genicular blocks (dexamethazone and lidocaine) — Genicular blocks were applied bilaterally by another physiatrist who was experienced in ultrasonographic (US) interventional procedures more than 5 years. Total of 6mL solution consisting of 0.5 mg/2mL dexamethazone and 4mL %1 lidocaine for three branches of genicular nerves (superomedial, superolateral and inferomedial branches) was divided into three branches for each knee. Total of 12 mL solution was applied for each patient.

SUMMARY:
Genicular nerve block (GNB) is a novel and promising interventional method for pain in knee osteoarthritis (KOA). However ,it contains afferent fibers that receive impulses from proprioceptive and deep sensory receptors located in the joint capsule, ligaments, muscles, tendons and periosteum. These proprioceptive stimuli are effective on joint position and biomechanics, protect the joint from injuries and help maintain balance. This study aims to evaluate Pproprioception and static balance after ultrasound-guided GNB in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Genicular nerve block (GNB) is a novel and promising interventional method for pain in knee osteoarthritis (KOA). However ,it contains afferent fibers that receive impulses from proprioceptive and deep sensory receptors located in the joint capsule, ligaments, muscles, tendons and periosteum. These proprioceptive stimuli are effective on joint position and biomechanics, protect the joint from injuries and help maintain balance. This study aims to evaluate Pproprioception and static balance after ultrasound-guided GNB in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic knee pain more than >3 according to visual analog scale (VAS) and difficulty in function more than 3 months
* Grade 2-3 KOA according to the Kellgren -Lawrence radiological grading system
* No significant improvement in response to conservative treatments such as analgesics and physiotherapy.

Exclusion Criteria:

* History of trauma, fractures, malignencies, surgery and inflammatory diseases of knee
* Limitation of range of motion in unilaterally and/or bilaterally in knee joint
* Allergies of pharmacological agents using during procedure (lidocaine)
* Presence of intra-articular or peri-articular injection such as hyaluronic acids, corticosteroids or collagen supplements at last 6 months
* Other neurologic or rheumatological conditions that may lead vertigo or vestibular disfunction or presence of impairment in proprioception such as polineuropathy
* Presence of diabetes mellitus due to risk of small fiber neuropathy
* Cognitive impairment and uncontrolled systemic conditions.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-14 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 24 hours
  Ten-cm VAS was used as a self-report measure for knee joint pain. Turkish Validity and Reliability of scale was published. 0 indicates no pain and 10 indicates unbearable pain. As it approaches 10, the pain becomes more severe.
HUR SmartBalance®: HUR SmartBalance® | 24 hours
  provides both balance assessments and rehabilitative training programs. Training programs are used in vertigo rehabilitation, balance training in mild gait disorders and fall prevention in elderly. Balance scores allow assessments and comparison in terms of static balance, proprioception disturbance, visual dependency and vestibular dominant proprioception . It consists of Balance Trainer, Support Rail, SmartBalance Software, Touchscreen Computer and Foam surface

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)